CLINICAL TRIAL: NCT01240421
Title: An Open-Label, Multi-Center, Expanded Access Program With Eribulin for the Treatment of Advanced Breast Cancer Refractory
Status: Approved for marketing | Type: Expanded Access
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: E7389-G000-398
Record Dates: First submitted 2010-10-01; First posted 2010-11-15 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic breast cancer with no other treatment options
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin

INTERVENTIONS:
Drug: Eribulin Mesylate — At a dose of 1.4 mg/m2 as a 2 to 5 minute intravenous bolus on Days 1 and 8 of a 21-day cycle.

SUMMARY:
This expanded access program is an open-label, multi-center study, which will consist of a PreTreatment Phase and a Treatment Phase. Patients with locally advanced or metastatic breast cancer who fulfill the eligibility criteria will be treated. The program will continue in each country until eribulin is approved, reimbursed and launched in that country, or termination of the program by the Sponsor.

ELIGIBILITY:
Key Inclusion Criteria:

* Patient's oncologist must have documented experience in a prior eribulin clinical trial
* Recurrent, locally advanced or metastatic breast cancer that has progressed on or after the last anti-cancer therapy
* Prior treatment with, ineligibility for, or commercial unavailability of each of the following therapies:

  1. Anthracyclines, taxanes, and capecitabine
  2. Ixabepilone, in countries where this agent is marketed
  3. Trastuzumab, for Her-2 positive disease
  4. Hormonal therapy, in hormone receptor-positive disease
  5. All other commercially available therapies, e.g. gemcitabine or vinorelbine, used for the treatment of advanced breast cancer (see NCCN guidelines)
* ECOG performance status greater than or equal to 2
* Adequate kidney function: serum creatinine less than or equal to 2.0 mg/dL or creatinine clearance greater than or equal to 40 mL/min
* Adequate bone marrow function: absolute neutrophil count greater than or equal to 1.5 x 10^9/L, hemoglobin greater than or equal to 10 g/dL (can be corrected by growth factor or transfusion), and platelet count greater than or equal to 100 x 10^9/L
* Adequate liver function: total bilirubin less than or equal to 1.5 x upper limit of normal (ULN), alkaline phosphatase, alanine aminotransferase, and aspartate aminotransferase less than or equal to 3 x ULN (or less than or equal to 5 x ULN in case of liver metastases). If alkaline phosphatase is greater than 3 x ULN (in absence of liver metastases) or greater than 5 x ULN (in presence of liver metastases) AND patient also is known to have bone metastases, the liver specific alkaline phosphatase must be used to assess liver function instead of total alkaline phosphatase
* Willing and able to comply with all aspects of the treatment protocol
* Provision of written informed consent
* Female, aged at least 18 years
* Patients of childbearing potential must agree to be abstinent or to use a highly effective method of contraception

Key Exclusion Criteria:

Eligibility for any other eribulin study open in the same region

* Existing anti-cancer therapy-related toxicities of grade 2 or more, except that alopecia and grade 2 neuropathy are acceptable
* History of congestive heart failure with New York Heart Association Classification greater than grade II, unstable angina, myocardial infarction within the past 6 months or serious cardiac arrhythmia
* Electrocardiogram with QTc interval of greater than or equal to 500 msec based upon Bazett's formula (QTcB)
* The Investigator believes the patient to be medically unfit to receive eribulin or unsuitable for any other reason
* Pregnancy (positive B-hCG test) or breastfeeding
* Hypersensitivity to eribulin or any of the excipients
* Brain or subdural metastases, unless local therapy has been completed and use of corticosteroids for this indication has been discontinued for at least 4 weeks before starting treatment in this protocol. Any signs (eg, radiologic) and/or symptoms of brain metastases must be stable for at least 4 weeks before starting the treatment protocol
* History of or concomitant medical condition that, in the opinion of the Investigator, would compromise the patient's ability to safely complete the treatment protocol
* Known human immunodeficiency virus positivity, as neutropenia caused by eribulin treatment may make such patients particularly susceptible to infection.
* Meningeal carcinomatosis
* Pulmonary lymphangitic involvement resulting in pulmonary dysfunction requiring active treatment, including use of oxygen
* Receipt of any of the following treatments within the specified period before the start of treatment: 1) Any investigational drug within 4 weeks; 2) Chemotherapy, radiation, biological or targeted therapy within 2 weeks; 3) Hormonal therapy within 1 week.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Dates: Start 2011-03; Primary Completion 2015-03 (Estimated); Study Completion 2014-11 (Estimated)

CONTACTS AND LOCATIONS:
Locations (14):
- Brussels, Belgium
- Canada (8):
  - Edmonton
  - London
  - Moncton
  - Montreal
  - Ottawa
  - Québec
  - Toronto
  - Vancouver
- France (5):
  - Besançon
  - Marseille
  - Paris
  - Saint-Cloud
  - Toulouse